CLINICAL TRIAL: NCT02278523
Title: The Respiratory Physiology Variation of COPD Patients in Inspiratory Muscle Training
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weiliang Wu, Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GuangzhouIRD; GuangzhouIRD (Other: GuangzhouIRD)
Record Dates: First submitted 2014-10-15; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory muscle training group (Experimental): COPD patient use Inspiratory muscle trainer (Threshold IMT®)
  Interventions: Device: Threshold IMT®
- control group (Active Comparator): normal volunteers use Inspiratory muscle trainer(Threshold IMT®)
  Interventions: Device: Threshold IMT®

INTERVENTIONS:
Device: Threshold IMT® — A device used to offer threshold load to inspiratory muscle
  Other Names: threshold inspiratory muscle trainer

SUMMARY:
Background：Respiratory muscle weakness is observed in chronic obstructive pulmonary disease(COPD) patients and contributes to hypercapnia, dyspnoea, nocturnal oxygen desaturation and reduced walking distance.During exercise it has been shown that diaphragm work is increased in COPD and COPD patients use a larger proportion of the maximal inspiratory pressure (MIP) than healthy subjects. This pattern of breathing is closely related to the dyspnoea sensation during exercise and might potentially induce respiratory muscle fatigue. Inspiratory muscle training(IMT) increases inspiratory muscle strength and endurance, and decreases dyspnoea.But the mechanism of IMT still lack of research.

Purpose：The experiment is aim to compare of the similarities and differences of transdiaphragmatic pressure by detecting the transdiaphragmatic pressure of COPD patients and healthy volunteers in different intensity of threshold load conditions. Thus investigate how inspiratory muscle training works or mechanism in lung rehabilitation programmes of COPD.And emerging the theoretical basis of inspiratory muscle training from respiratory physiological mechanism.

DETAILED DESCRIPTION:
Subjects:

COPD group ( experimental group ) Ten subjects with moderate COPD were will be recruited from the investigators outpatient clinic for the study. According to the criteria of the American Thoracic Society (ATS), COPD is defined as postbronchodilator forced expiratory volume in 1 second (FEV1) of 30% to 79% of the predicted value and a ratio of FEV1 to forced vital capacity (FVC) ,70%.

Inclusion criteria:(1)Severe and very severe COPD (postbronchodilator FEV1/FVC under 70% and FEV1 under 50% of the predicted value;(2)Inspiratory muscle weakness（Maximal Inspiratory Pressure under 60cmH2O（centimeter water column）.(3) bronchial dilation test(BDT) negative.(4) Exclusion of other cardiopulmonary diseases.

Exclusion criterion:(1)Suffer from acute exacerbation less than 4 weeks.(2) Intravenous or oral corticosteroids in 4 weeks.(3) With other heart, lung and brain disorders.(4) With poor compliance.

Healthy volunteers group (control group ) Inclusion criteria:(1) Normal lung function(FEV1/FVC above 70% and FEV1 above 50% of the predicted value); (2)Without inspiratory muscle weakness（Maximal Inspiratory Pressure above 60cmH2O）(3) without nervous system and respiratory diseases.

Experimental methods : prospective randomized controlled trial（RCT）

1. record the information of the subjects: sexuality, age ( years ), height ( cm), weight ( kg ), BMI ;
2. Pulmonary function tests:forced expiratory volume in 1 second（FEV1）, FEV1 of the predicted value (FEV1/Pred%), forced vital capacity (FVC), FVC of the predicted value (FVC/Pred%), a ratio of FEV1 to forced vital capacity (FEV1/FVC%).
3. Synchronous record:mouth pressure ( Pm ), esophageal pressure ( Peso ), intragastric pressure ( Pgas ),transdiaphragmatic pressure ( Pdi ), flow ( flow ), tidal volume ( volume ), Five lead diaphragmatic electromyography of the esophagus ( electromyography diaphragm （EMGdi1, EMGdi2, EMGdi3, EMGdi4, EMGdi5 )）.
4. Measure the maximal inspiratory pressure, records of maximum transdiaphragmatic pressure and maximum diaphragmatic electromyography simultaneously.

Subjects suffer from different level of threshold load generated by threshold loading device. Detecting the pressure and electrical while adjust the load to 30%,40%,50%,60%,70%,80% of the MIP respectively. The change from baseline in transdiaphragmatic pressure will be detect in each level of load.

ELIGIBILITY:
Inclusion Criteria:

* Severe and very severe COPD (postbronchodilator FEV1/FVC under 70% and FEV1 under 50% of the predicted value
* Inspiratory muscle weakness（Maximal Inspiratory Pressure under 60cmH2O.
* Bronchial dilation test(BDT) negative.
* Exclusion of other cardiopulmonary diseases.

Exclusion Criteria:

* Suffer from acute exacerbation less than 4 weeks.
* Intravenous or oral corticosteroids in 4 weeks.
* With other heart, lung and brain disorders.
* With poor compliance.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Transdiaphragmatic pressure | half an hour
  measure the transdiaphragmatic pressure while spontaneous breathing

CONTACTS AND LOCATIONS:
Overall Officials: Chen Rongchang, Master, Study Chair — Guangzhou Institude of Respiratory Disease
Locations (1):
- Respiratory muscle training device, Guangzhou, Guangdong, China